CLINICAL TRIAL: NCT03181893
Title: A PHASE 2 DOUBLE-BLIND, RANDOMIZED, PLACEBO-CONTROLLED STUDY TO EVALUATE THE EFFICACY, SAFETY, AND TOLERABILITY OF PF-06823859 IN ADULT SUBJECTS WITH DERMATOMYOSITIS
Brief Title: A Study In Adults With Moderate To Severe Dermatomyositis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: C0251002; 2020-004228-41 (EudraCT Number)
Record Dates: First submitted 2017-06-05; First posted 2017-06-09 (Actual); Results first posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Dermatomyositis
MeSH Terms: conditions — Dermatomyositis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo ARM (Placebo Comparator)
  Interventions: Drug: Placebo Arm
- PF-06823859 ARM high (Experimental)
  Interventions: Drug: PF-06823859 high
- PF-06823859 ARM low (Experimental)
  Interventions: Drug: PF-06823859 low

INTERVENTIONS:
Drug: PF-06823859 low — A humanized immunoglobulin neutralizing antibody
  Arms: PF-06823859 ARM low
Drug: Placebo Arm — Placebo contains histidine, sucrose, PS80, ethylene diamine, and triacetic acid
  Arms: Placebo ARM
Drug: PF-06823859 high — A humanized immunoglobulin neutralizing antibody
  Arms: PF-06823859 ARM high

SUMMARY:
A Study looking at Investigational drug and Placebo administered to adult Patients with moderate to severe Dermatomyositis

ELIGIBILITY:
Inclusion Criteria for Patients with Skin Predominant Activity:

* Must have CDASI Activity score of greater than or equal to 14, and have failed at least 1 standard of care systemic treatment, (eg, corticosteroids).
* Confirmation of DM by the investigator and two of the following:

  1. Gottron's papules;
  2. Gottron's sign;
  3. Heliotrope eruption;
  4. Nailfold changes, (dilated capillary loops, capillary dropout, cuticular hypertrophy and/or rugged cuticles;
  5. Photodistributed violaceous erythema, (skin that is exposed to sunlight and appears purplish/reddish, and patchy in appearance;
  6. Positive DM serology -
* Post DM diagnosis; standard of care workup for DM must have been completed prior to entry into this research study.
* Willing to provide 8 biopsies during the course of the research study

Inclusion Criteria for Patients with Muscle Predominant Activity:

* MMT-8 ≤136/150 and PhGA, VAS ≥3 cm (0-10 cm) by visual analog scale (VAS)
* Sum of PhGA, VAS, PtGA, and extramuscular global assessment VAS scores is ≥10 cm (0-10 cm) VAS for each.

  * Participant has failed at least two or more adequate courses of an immunosuppressive agent or immunomodulatory agent, including IVIG, at a dose known to be effective for rheumatologic diseases.

Exclusion Criteria for Patients with Skin Predominant Activity:

* Investigator site staff or members of their family.
* Acute and Chronic present medical conditions
* Intake of greater than 15 mg of prednisone or equivalent per day
* Pregnant or breastfeeding females. Fertile men and women who will not comply with the use of 2 effective birth control methods as per the research protocol
* Have required management of acute or chronic infections
* Have pre existing demyelinating disorder such as multiple sclerosis, or other severe neurological deficits.
* Clinically significant lab abnormalities
* Any health condition that may be worsened by immunosuppression

Exclusion Criteria for Patients with Muscle Predominant Activity:

Similar to patients with skin predominant activity; Intake of >20 mg oral prednisone/day, or equivalent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (40):
- United States (34):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Arizona Research Pharmacy, Phoenix, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - Attune Health Research Inc., Beverly Hills, California
  - Freidenrich Center for Translational Research at Stanford University, Palo Alto, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - University Of Miami Hospital, Miami, Florida
  - University of Miami Hospital Clinical Translational Research Site (Infusion site), Miami, Florida
  - KU Clinical Research Center - Clinical and Translational Science Unit (CTSU), Fairway, Kansas
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Brigham and Women's Hospital - ACC, Boston, Massachusetts
  - Brigham and Women's Hospital - CTC, Boston, Massachusetts
  - Brigham and Women's Hospital - CTH, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Clinical Research Unit (CRU), Minneapolis, Minnesota
  - Department of Medicine Division of Rheumatic and Autoimmune Disease, Minneapolis, Minnesota
  - Lillehei Clinical Research Unit (LCRU), Minneapolis, Minnesota
  - University of Minnesota Health Rheumatology Clinic, Minneapolis, Minnesota
  - University of Minnesota, Department of Dermatology, Minneapolis, Minnesota
  - Center for Outpatient Health, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - New York University School of Medicine, New York, New York
  - NYU Langone Health Clinical Research Center, New York, New York
  - Mount Sinai Doctors Dermatology, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - OHSU, Center for Health and Healing CHH2, Portland, Oregon
  - Oregon Clinical & Translational Research Institute, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Utah MidValley Dermatology, Murray, Utah
  - Center for Clinical & Translational Science, Salt Lake City, Utah
- Universitaetsklinikum Tuebingen, Tübingen, Germany
- University of Debrecen, Debrecen, Hajdú-Bihar, Hungary
- Poland (2):
  - Nova Reuma spolka partnerska, Bialystok
  - Centrum Medyczne Plejady, Krakow
- Spain (2):
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Quiron Infanta Luisa, Seville

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Fiorentino D, Mangold AR, Werth VP, Christopher-Stine L, Femia A, Chu M, Musiek ACM, Sluzevich JC, Graham LV, Fernandez AP, Aggarwal R, Rieger K, Page KM, Li X, Hyde C, Rath N, Sloan A, Oemar B, Banerjee A, Salganik M, Banfield C, Neelakantan S, Beebe JS, Vincent MS, Peeva E, Vleugels RA. Efficacy, safety, and target engagement of dazukibart, an IFNbeta specific monoclonal antibody, in adults with dermatomyositis: a multicentre, double-blind, randomised, placebo-controlled, phase 2 trial. Lancet. 2025 Jan 11;405(10473):137-146. doi: 10.1016/S0140-6736(24)02071-3. PMID 39798982
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C0251002

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 75 participants were randomized at 19 centers in 5 countries: 32, 9, 16 and 18 participants were treated in Stage 1, Stage 2, Amended Stage 2 and Stage 3, respectively.
  A fixed sequence design with crossover at Week 12 was employed in Amended Stage 2 and Stage 3 to provide all participants with the opportunity to receive active drug during the treatment period.
Groups:
- (Stage 1) Placebo: Participants in this group were randomized to receive placebo on Day 1, Week 4, and Week 8 in Stage 1 After week 12, participants went into a follow up period.
- (Stage 1) PF-06823859 600 mg Intravenous (IV): Participants in this group were randomized to receive PF-06823859 600 mg on Day 1, Week 4, and Week 8 in Stage 1. After week 12, participants went into a follow up period.
- (Stage 2) Placebo: Participants in this group were randomized to receive placebo on Day 1, Week 4, and Week 8 in Stage 2. After week 12, participants went into a follow up period.
- (Stage 2) PF-06823859 150 mg IV: Participants in this group were randomized to receive PF-06823859 150 mg on Day 1, Week 4, and Week 8. After week 12, participants went into a follow up period.
- (Stage 2) PF-06823859 600 mg IV: Dosing occurred Day 1, Week 4, and Week 8. After week 12, participants went into a follow-up period.
- (Amended Stage 2) Placebo Then Switched to PF-06823859 150 mg IV at Week 12: Dosing occurred Day 1, Weeks 4, 8, 12, 16, 20. At Week 24, participants then entered a 4-month follow-up period or rolled over to the long-term extension study.
- (Amended Stage 2) Placebo Then Switched to PF-06823859 600 mg IV at Week 12: Dosing occurred on Day 1, Weeks 4, 8, 12, 16, 20. At Week 24, participants then entered a 4-month follow-up period or rolled over to the long-term extension study.
- (Amended Stage 2) PF-06823859 150 mg IV Then Switched to Placebo at Week 12: Dosing occurred Day 1, Weeks 4, 8, 12, 16 and 20. At Week 24, participants then entered a 4-month follow-up period or rolled over to the long-term extension study.
- (Amended Stage 2) PF-06823859 600 mg IV Then Switched to Placebo at Week 12: Dosing occurred Day 1, Weeks 4, 8, 12, 16, and 20. At Week 24, participants then entered a 4-month follow-up period or rolled over to the long-term extension study.
- (Stage 3) Placebo Then Switched to PF-06823859 600 mg IV at Week 12: Dosing occurred Day 1, Weeks 4, 8, 12, 16, 20. At Week 24, participants entered a 4-month follow-up period or rolled over to the long-term extension study.
- (Stage 3) PF-06823859 600 mg IV Then Switched to Placebo at Week 12: Dosing occurred Day 1, Weeks 4, 8, 12, 16, and 20. At Week 24, participants entered a 4-month follow-up period or rolled over to the long-term extension study.
Period: Baseline to Week 12 (All Stages)
Arm/Group | (Stage 1) Placebo | (Stage 1) PF-06823859 600 mg Intravenous (IV) | (Stage 2) Placebo | (Stage 2) PF-06823859 150 mg IV | (Stage 2) PF-06823859 600 mg IV | (Amended Stage 2) Placebo Then Switched to PF-06823859 150 mg IV at Week 12 | (Amended Stage 2) Placebo Then Switched to PF-06823859 600 mg IV at Week 12 | (Amended Stage 2) PF-06823859 150 mg IV Then Switched to Placebo at Week 12 | (Amended Stage 2) PF-06823859 600 mg IV Then Switched to Placebo at Week 12 | (Stage 3) Placebo Then Switched to PF-06823859 600 mg IV at Week 12 | (Stage 3) PF-06823859 600 mg IV Then Switched to Placebo at Week 12
Started | 10 | 22 | 1 | 5 | 3 | 2 | 1 | 10 | 3 | 9 | 9
Completed | 9 | 20 | 1 | 5 | 3 | 2 | 1 | 10 | 3 | 9 | 9
Not Completed | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Weeks 12-24 (Amended Stage 2, Stage 3)
Arm/Group | (Stage 1) Placebo | (Stage 1) PF-06823859 600 mg Intravenous (IV) | (Stage 2) Placebo | (Stage 2) PF-06823859 150 mg IV | (Stage 2) PF-06823859 600 mg IV | (Amended Stage 2) Placebo Then Switched to PF-06823859 150 mg IV at Week 12 | (Amended Stage 2) Placebo Then Switched to PF-06823859 600 mg IV at Week 12 | (Amended Stage 2) PF-06823859 150 mg IV Then Switched to Placebo at Week 12 | (Amended Stage 2) PF-06823859 600 mg IV Then Switched to Placebo at Week 12 | (Stage 3) Placebo Then Switched to PF-06823859 600 mg IV at Week 12 | (Stage 3) PF-06823859 600 mg IV Then Switched to Placebo at Week 12
Started (Participants from Stage 1 or Stage 2 did not participate in the treatment switch from Week 12 to 24. Therefore, not applicable for this period.) | 0 (Not applicable for this period.) | 0 (Not applicable for this period.) | 0 (Not applicable for this period.) | 0 (Not applicable for this period.) | 0 (Not applicable for this period.) | 2 | 1 | 10 | 3 | 9 | 9
Completed | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 9 | 2 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis population included all participants who had received at least 1 dose of study drug or placebo.
Groups:
- (Stage 1) Placebo; (Stage 2) Placebo: Participants in this group were randomized to receive placebo on Day 1, Week 4, and Week 8. After week 12, participants went into a follow up period.
- (Stage 1) PF-06823859 600 mg Intravenous (IV): Participants in this group were randomized to receive PF-06823859 600 mg on Day 1, Week 4, and Week 8.
  After week 12, participants went into a follow up period.
- (Stage 2) PF-06823859 150 mg IV: Participants in this group were randomized to receive PF-06823859 150 mg on Day 1, Week 4, and Week 8 After week 12, participants went into a follow up period.
- Total: Total of all reporting groups
Arm/Group | (Stage 1) Placebo | (Stage 1) PF-06823859 600 mg Intravenous (IV) | (Stage 2) Placebo | (Stage 2) PF-06823859 150 mg IV | (Stage 2) PF-06823859 600 mg IV | (Amended Stage 2) Placebo Then Switched to PF-06823859 150 mg IV at Week 12 | (Amended Stage 2) Placebo Then Switched to PF-06823859 600 mg IV at Week 12 | (Amended Stage 2) PF-06823859 150 mg IV Then Switched to Placebo at Week 12 | (Amended Stage 2) PF-06823859 600 mg IV Then Switched to Placebo at Week 12 | (Stage 3) Placebo Then Switched to PF-06823859 600 mg IV at Week 12 | (Stage 3) PF-06823859 600 mg IV Then Switched to Placebo at Week 12 | Total
Number analyzed (Participants) | 10 | 22 | 1 | 5 | 3 | 2 | 1 | 10 | 3 | 9 | 9 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.20 (14.054) | 54.41 (13.154) | 42.00 | 51.60 (15.726) | 45.67 (23.714) | 64.00 (1.414) | 44 | 53.90 (10.999) | 47.00 (13.115) | 47.44 (12.126) | 42.44 (16.697) | 50.63 (13.793)
Age, Customized [Count of Participants; unit: Participants]
  18-64 Years | 8 | 18 | 1 | 4 | 2 | 1 | 1 | 8 | 3 | 8 | 8 | 62
  65-84 Years | 2 | 4 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 1 | 1 | 13
  >=85 Years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 20 | 1 | 5 | 3 | 2 | 1 | 10 | 2 | 6 | 7 | 66
  Male | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 3 | 2 | 13
  Not Hispanic or Latino | 8 | 20 | 0 | 5 | 2 | 2 | 1 | 9 | 2 | 6 | 7 | 62
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 9 | 20 | 1 | 5 | 3 | 2 | 1 | 9 | 3 | 8 | 8 | 69
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Multiracial | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Not reported | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Cutaneous Dermatomyositis Disease Area and Severity Index (CDASI) Activity Score at Week 12 (Stage 1, Stage 2 and Amended Stage 2)
Description: The treatment effect was defined as the difference (mean chg from baseline at Week12 in the active treatment group minus that in the placebo group) in the mean change of CDASI activity score from baseline at Week 12. The score (range: 0-100) consists of the extent score (ES), Gottorn hands score (GHS), peringual score (PS) and allopecia score (AS). ES (range: 0-90) was obtained by summing up scores for the total erythema (ER [0-45], redness of the skin or mucous membranes), scaling (SC [0-30], peeling of the skin) and erosion/ulceration (EU [0-15], presence of the deeper wound). Total ER, SC and EU scores were calculated as a sum of the contributions from 15 individual areas of the body. GHS characterizes papules (swellings) on hand and is a sum of the papule's characterization score (0-6) and ulceration score (0-1). PS (0-2) characterizes abnormalities around nails. The AS (0-1) characterizes hair loss. Higher scores indicate greater disease severity.
Time Frame: Baseline and Week 12
Population: The Full Analysis Set (FAS) in Stage 1, Stage 2, and Amended Stage 2 included all participants who received at least 1 dose of randomized treatment in in Stage 1, Stage 2, or Amended Stage 2.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- PF-06823859 600 mg IV (Stage 1): Participants were randomized to receive PF-06823859 600 mg on Day 1, Week 4, and Week 8 in Stage 1.
Arm/Group | (Stage 1) Placebo | PF-06823859 600 mg IV (Stage 1) | (Stage 2) Placebo | (Stage 2) PF-06823859 150 mg IV | (Stage 2) PF-06823859 600 mg IV | (Amended Stage 2) Placebo Then Switched to PF-06823859 150 mg IV at Week 12 | (Amended Stage 2) Placebo Then Switched to PF-06823859 600 mg IV at Week 12 | (Amended Stage 2) PF-06823859 150 mg IV Then Switched to Placebo at Week 12 | (Amended Stage 2) PF-06823859 600 mg IV Then Switched to Placebo at Week 12
Number analyzed (Participants) | 9 | 21 | 1 | 5 | 3 | 2 | 1 | 10 | 3
Units on a scale | -3.44 (5.270) | -19.62 (9.140) | 5.00 | -17.40 (9.290) | -26.00 (7.937) | -3.00 (8.485) | 3.00 | -16.40 (5.835) | -15.33 (6.028)
Statistical Analysis 1: Comparison: (Stage 1) Placebo vs PF-06823859 600 mg IV (Stage 1); Test type: Other; p < 0.0001, LANCOVA-P model; Mean Difference (Final Values) = -14.82, 90% CI 2-sided [-20.26 to -9.37], Standard Error of Mean 3.183

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAE) (Stage 3)
Description: Adverse event (AE) was any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. SAE was any untoward medical occurrence that at any dose resulted in any of following outcomes/deemed significant for any other reason: death; initial /prolonged inpatient hospitalization; life-threatening; persistent or significant disability/incapacity; congenital anomaly/birth defect and suspected transmission via a Pfizer product of an infectious agent, pathogenic or non-pathogenic. AEs included both serious (if occurred) and all non-serious adverse events. TEAEs are events between first dose of study drug and up to Week 40 that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Up to Week 40
Population: The safety analysis set in Stage 3 (SAS3) included all participants who received at least 1 dose of randomized treatment in Stage 3.
Measure: Count of Participants; unit: Participants
Arm/Group | (Stage 3) Placebo Then Switched to PF-06823859 600 mg IV at Week 12 | (Stage 3) PF-06823859 600 mg IV Then Switched to Placebo at Week 12
Number analyzed (Participants) | 9 | 9
Participants
  TEAEs | 7 | 8
  SAEs | 0 | 2

3. Primary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities (Stage 3)
Description: Hemoglobin(HGB),hematocrit,erythrocytes(ery.),HDL cholesterol(chl.)<0.8*lower limit of normal(LLN);reticulocytes (ret.), ret./ery.(%)<0.5*LLN,>1.5*upper limit of normal (ULN);ery. mean corpuscular(EMC) volume,EMC HGB concentration,potassium,chloride,calcium,bicarbonate<0.9*LLN,>1.1*ULN;platelets<0.5*LLN,>1.75*ULN; leukocytes(leu.),glucose<0.6*LLN,>1.5*ULN;lymphocytes(lym.), lym./leu.(%),neutrophils (neu.), neu./leu.(%), protein,albumin<0.8*LLN,>1.2*ULN;basophils(bas.), bas./leu.(%), eosinophils(eos.), eos./leu., monocytes(mon.), mon./leu.(%), urate>1.2*ULN;bilirubin (total, direct,indirect)>1.5*ULN;aspartate/alanine aminotransferase,gamma glutamyl transferase,lactate dehydrogenase,alkaline phosphatase>3.0*ULN;urea nitrogen,creatinine,triglycerides, chl.>1.3*ULN; sodium <0.95*LLN,>1.05*ULN; creatine kinase >2.0*ULN;Urine: pH<4.5,>8;glucose, ketones,protein, HGB,urobilinogen,bilirubin,nitrite,leukocyte esterase>=1;ery., leu.>= 20;hyaline casts>1;bacteria>20.
Time Frame: Up to Week 40
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | (Stage 3) Placebo Then Switched to PF-06823859 600 mg IV at Week 12 | (Stage 3) PF-06823859 600 mg IV Then Switched to Placebo at Week 12
Number analyzed (Participants) | 9 | 9
Participants | 0 | 1

4. Primary Outcome: Number of Participants With Vital Sign Abnormalities (Stage 3)
Description: Abnormality in vital signs: Sitting pulse rate <40 beats per minute (bpm) to >120 bpm, sitting diastolic blood pressure (DBP) < 50 millimeter of mercury (mmHg), sitting systolic blood pressure (SBP) <90 mmHg.
Time Frame: Baseline up to Week 40
Population: The SAS3 included all participants who received at least 1 dose of randomized treatment in Stage 3.
Measure: Count of Participants; unit: Participants
Arm/Group | (Stage 3) Placebo Then Switched to PF-06823859 600 mg IV at Week 12 | (Stage 3) PF-06823859 600 mg IV Then Switched to Placebo at Week 12
Number analyzed (Participants) | 9 | 9
Participants
  Sitting SBP Value <90 mmHg | 0 | 0
  Sitting DBP Value <50 mmHg | 0 | 0
  Sitting Pulse Rate Value <40 bpm | 0 | 0
  Sitting Pulse Rate Value >120 bpm | 0 | 0

5. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities (Stage 3)
Description: ECG abnormalities criteria included: 1) QTc interval adjusted according to Fridericia formula (QTcF) (msec): >450, >480, >500, increase from baseline >=30, increase from baseline >=60; 2) Pulse rate (PR) (msec): >=300, change from baseline (Chg) >=25% or 50%; 3) QT (msec): >=500; 4) QRS (msec): >=200, Chg >=25% or 50%. Categories, with at least 1 participant having ECG abnormality in any of the reporting arms, were reported in this outcome measure.
Time Frame: Baseline up to Week 40
Population: The SAS3 included all participants who received at least 1 dose of randomized treatment in Stage 3.
Measure: Count of Participants; unit: Participants
Arm/Group | (Stage 3) Placebo Then Switched to PF-06823859 600 mg IV at Week 12 | (Stage 3) PF-06823859 600 mg IV Then Switched to Placebo at Week 12
Number analyzed (Participants) | 9 | 9
Participants
  PR Interval Aggregate Value >=300 msec | 0 | 0
  QRS Duration Aggregate Value >=200 msec | 0 | 0
  QT Interval Aggregate Value >=500 msec | 0 | 0
  QTcF Interval Aggregate 450<=Value<480 msec | 0 | 1
  QTcF Interval Aggregate 480<=Value<500 msec | 1 | 0
  QTcF Interval Aggregate Value >=500 msec | 0 | 0
  PR %Chg >=25% or >=50% | 0 | 0
  QRS Duration %Chg >=25% or >=50% | 0 | 0
  30<=QTcF Chg (msec)<60 | 0 | 0
  QTcF Chg (msec) >=60 | 0 | 1

6. Secondary Outcome: Number of Participants With TEAEs and SAEs (Stage 1 and Stage 2)
Description: AE was any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. SAE was any untoward medical occurrence that at any dose resulted in any of following outcomes/deemed significant for any other reason: death; initial /prolonged inpatient hospitalization; life-threatening; persistent or significant disability/incapacity; congenital anomaly/birth defect and suspected transmission via a Pfizer product of an infectious agent, pathogenic or non-pathogenic. AEs included both serious (if occurred) and all non-serious adverse events. TEAEs are events between first dose of study drug and up to Week 28 that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Up to Week 28
Population: The safety analysis set in Stage 1 (SAS1) and safety analysis set in Stage 2 (SAS2) included all participants who received at least 1 dose of randomized treatment in Stage 1 and Stage 2, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | (Stage 1) Placebo | PF-06823859 600 mg IV (Stage 1) | (Stage 2) Placebo | (Stage 2) PF-06823859 150 mg IV | (Stage 2) PF-06823859 600 mg IV
Number analyzed (Participants) | 10 | 22 | 1 | 5 | 3
Participants
  TEAEs | 8 | 20 | 1 | 5 | 3
  SAEs | 1 | 2 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With TEAEs and SAEs (Amended Stage 2)
Description: AE was any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. SAE was any untoward medical occurrence that at any dose resulted in any of following outcomes/deemed significant for any other reason: death; initial /prolonged inpatient hospitalization; life-threatening; persistent or significant disability/incapacity; congenital anomaly/birth defect and suspected transmission via a Pfizer product of an infectious agent, pathogenic or non-pathogenic. AEs included both serious (if occurred) and all non-serious adverse events. TEAEs are events between first dose of study drug and up to Week 40 that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Up to Week 40
Population: The safety analysis set in Amended Stage 2 (SASA2) includes all participants who received at least one dose of randomized treatment in Amended Stage 2.
Measure: Count of Participants; unit: Participants
Arm/Group | (Amended Stage 2) Placebo Then Switched to PF-06823859 150 mg IV at Week 12 | (Amended Stage 2) Placebo Then Switched to PF-06823859 600 mg IV at Week 12 | (Amended Stage 2) PF-06823859 150 mg IV Then Switched to Placebo at Week 12 | (Amended Stage 2) PF-06823859 600 mg IV Then Switched to Placebo at Week 12
Number analyzed (Participants) | 2 | 1 | 10 | 3
Participants
  TEAEs | 1 | 1 | 8 | 3
  SAEs | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities (Stage 1 and Stage 2)
Description: HGB,hematocrit,ery.,HDL chl.<0.8*LLN;ret., ret./ery. (%)<0.5*LLN,>1.5*ULN;EMC volume,EMC HGB,EMC HGB concentration,potassium,chloride,calcium,bicarbonate<0.9*LLN,>1.1*ULN;platelets<0.5*LLN,>1.75*ULN;leu.,glucose<0.6*LLN,>1.5*ULN;lym., lym./leu.(%), neu., neu./leu. (%), protein,albumin <0.8*LLN,>1.2*ULN;bas., bas./leu.(%), eos., eos./leu., mon., mon./leu.(%), urate >1.2*ULN;bilirubin (total, direct, indirect)>1.5*ULN;aspartate/alanine aminotransferase, gamma glutamyl transferase, lactate dehydrogenase, alkaline phosphatase>3.0*ULN;urea nitrogen, creatinine, triglycerides, chl.>1.3*ULN; sodium <0.95*LLN,>1.05*ULN; creatine kinase >2.0*ULN;Urine: pH<4.5,>8;glucose, ketones, protein, HGB, urobilinogen,bilirubin,nitrite,leukocyte esterase>=1;ery., leu.>= 20;hyaline casts>1;bacteria>20. Clinical significance of laboratory parameters was determined at the investigator's discretion.
Time Frame: Up to Week 28
Population: The SAS1 and SAS2 included all participants who received at least 1 dose of randomized treatment in Stage 1 and Stage 2, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | (Stage 1) Placebo | PF-06823859 600 mg IV (Stage 1) | (Stage 2) Placebo | (Stage 2) PF-06823859 150 mg IV | (Stage 2) PF-06823859 600 mg IV
Number analyzed (Participants) | 10 | 22 | 1 | 5 | 3
Participants | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities (Amended Stage 2)
Description: as for outcome 8
Time Frame: Up to Week 40
Population: The SASA2 includes all participants who received at least one dose of randomized treatment in Amended Stage 2.
Measure: Count of Participants; unit: Participants
Arm/Group | (Amended Stage 2) Placebo Then Switched to PF-06823859 150 mg IV at Week 12 | (Amended Stage 2) Placebo Then Switched to PF-06823859 600 mg IV at Week 12 | (Amended Stage 2) PF-06823859 150 mg IV Then Switched to Placebo at Week 12 | (Amended Stage 2) PF-06823859 600 mg IV Then Switched to Placebo at Week 12
Number analyzed (Participants) | 2 | 1 | 10 | 3
Participants | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Vital Sign Abnormalities (Stage 1 and Stage 2)
Description: Abnormality in vital signs: Sitting pulse rate <40 bpm to >120 bpm, sitting DBP < 50 mmHg, sitting SBP <90 mmHg.
Time Frame: Up to Week 28
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | (Stage 1) Placebo | PF-06823859 600 mg IV (Stage 1) | (Stage 2) Placebo | (Stage 2) PF-06823859 150 mg IV | (Stage 2) PF-06823859 600 mg IV
Number analyzed (Participants) | 10 | 22 | 1 | 5 | 3
Participants
  Sitting SBP Value <90 mmHg | 0 | 1 | 0 | 0 | 0
  Sitting DBP Value <50 mmHg | 0 | 0 | 0 | 0 | 0
  Sitting Pulse Rate Value <40 bpm | 0 | 0 | 0 | 0 | 0
  Sitting Pulse Rate Value >120 bpm | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Vital Sign Abnormalities (Amended Stage 2)
Description: Abnormality in vital signs: Sitting pulse rate <40 bpm to >120 bpm, sitting DBP < 50 mmHg, sitting SBP <90 mmHg.
Time Frame: Up to Week 40
Population: The SASA2 includes all participants who received at least one dose of randomized treatment in Amended Stage 2.
Measure: Count of Participants; unit: Participants
Arm/Group | (Amended Stage 2) Placebo Then Switched to PF-06823859 150 mg IV at Week 12 | (Amended Stage 2) Placebo Then Switched to PF-06823859 600 mg IV at Week 12 | (Amended Stage 2) PF-06823859 150 mg IV Then Switched to Placebo at Week 12 | (Amended Stage 2) PF-06823859 600 mg IV Then Switched to Placebo at Week 12
Number analyzed (Participants) | 2 | 1 | 10 | 3
Participants
  Sitting SBP Value <90 mmHg | 0 | 0 | 0 | 0
  Sitting DBP Value <50 mmHg | 0 | 0 | 0 | 0
  Sitting Pulse Rate Value <40 bpm | 0 | 0 | 0 | 0
  Sitting Pulse Rate Value >120 bpm | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With ECG Abnormalities (Stage 1 and Stage 2)
Description: as for outcome 5
Time Frame: Up to Week 28
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | (Stage 1) Placebo | PF-06823859 600 mg IV (Stage 1) | (Stage 2) Placebo | (Stage 2) PF-06823859 150 mg IV | (Stage 2) PF-06823859 600 mg IV
Number analyzed (Participants) | 10 | 22 | 1 | 5 | 3
Participants
  PR Interval Aggregate Value >=300 msec | 0 | 0 | 0 | 0 | 0
  QRS Duration Aggregate Value >=200 msec | 0 | 0 | 0 | 0 | 0
  QT Interval Aggregate Value >=500 msec | 0 | 0 | 0 | 0 | 0
  QTcF Interval Aggregate 450<=Value<480 msec | 3 | 1 | 0 | 1 | 0
  QTcF Interval Aggregate 480<=Value<500 msec | 0 | 0 | 0 | 0 | 0
  QTcF Interval Aggregate Value >=500 msec | 0 | 1 | 0 | 0 | 0
  PR %Chg >=25% or >=50% | 0 | 0 | 0 | 0 | 0
  QRS Duration %Chg >=25% or >=50% | 0 | 0 | 0 | 0 | 0
  30<=QTcF Chg (msec)<60 | 0 | 0 | 0 | 0 | 0
  QTcF Chg (msec) >=60 | 0 | 1 | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With ECG Abnormalities (Amended Stage 2)
Description: as for outcome 5
Time Frame: Up to Week 40
Population: The SASA2 includes all participants who received at least one dose of randomized treatment in Amended Stage 2.
Measure: Count of Participants; unit: Participants
Arm/Group | (Amended Stage 2) Placebo Then Switched to PF-06823859 150 mg IV at Week 12 | (Amended Stage 2) Placebo Then Switched to PF-06823859 600 mg IV at Week 12 | (Amended Stage 2) PF-06823859 150 mg IV Then Switched to Placebo at Week 12 | (Amended Stage 2) PF-06823859 600 mg IV Then Switched to Placebo at Week 12
Number analyzed (Participants) | 2 | 1 | 10 | 3
Participants
  PR Interval Aggregate Value >=300 msec | 0 | 0 | 0 | 0
  QRS Duration Aggregate Value >=200 msec | 0 | 0 | 0 | 0
  QT Interval Aggregate Value >=500 msec | 0 | 0 | 0 | 0
  QTcF Interval Aggregate 450<=Value<480 msec | 1 | 0 | 3 | 0
  QTcF Interval Aggregate 480<=Value<500 msec | 0 | 0 | 0 | 0
  QTcF Interval Aggregate Value >=500 msec | 0 | 0 | 0 | 0
  PR %Chg >=25% or >=50% | 0 | 0 | 0 | 0
  QRS Duration %Chg >=25% or >=50% | 0 | 0 | 0 | 0
  30<=QTcF Chg (msec)<60 | 1 | 0 | 1 | 0
  QTcF Chg (msec) >=60 | 0 | 0 | 0 | 0

14. Secondary Outcome: Change From Baseline in CDASI Activity Score at at All Scheduled Timepoints Through Week 12 (Stage 1, Stage 2 and Amended Stage 2)
Description: The treatment effect was defined as the difference (mean change from baseline at Weeks 1, 4, 8 in the active treatment group minus the mean change from baseline at Weeks 1, 4, 8 in the placebo group) in the mean change of CDASI activity score from baseline at scheduled timepoints. The score (range: 0-100) consists of the ES, GHS, PS and AS. ES (range: 0-90) was obtained by summing up scores for the total erythema (ER [0-45], redness of the skin or mucous membranes), scaling (SC [0-30], peeling of the skin) and erosion/ulceration (EU [0-15], presence of the deeper wound). Total ER, SC and EU scores were calculated as a sum of the contributions from 15 individual areas of the body. GHS characterizes papules (swellings) on hand and is a sum of the papule's characterization score (0-6) and ulceration score (0-1). PS (0-2) characterizes abnormalities around nails. The AS (0-1) characterizes hair loss. Higher scores indicate greater disease severity.
Time Frame: Baseline, Week 1, Week 4, and Week 8 (except for Week 12 which is a primary outcome measure)
Population: The FAS in Stage 1, Stage 2, and Amended Stage 2 included all participants who received at least 1 dose of randomized treatment in in Stage 1, Stage 2, or Amended Stage 2.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | (Stage 1) Placebo | PF-06823859 600 mg IV (Stage 1) | (Stage 2) Placebo | (Stage 2) PF-06823859 150 mg IV | (Stage 2) PF-06823859 600 mg IV | (Amended Stage 2) Placebo Then Switched to PF-06823859 150 mg IV at Week 12 | (Amended Stage 2) Placebo Then Switched to PF-06823859 600 mg IV at Week 12 | (Amended Stage 2) PF-06823859 150 mg IV Then Switched to Placebo at Week 12 | (Amended Stage 2) PF-06823859 600 mg IV Then Switched to Placebo at Week 12
Number analyzed (Participants) | 10 | 21 | 1 | 5 | 3 | 2 | 1 | 10 | 3
Units on a scale
  Week 1 | -2.60 (4.326) | -19.62 (9.140) | 1.00 | -9.80 (12.174) | -2.33 (1.528) | -6.50 (6.364) | 0.00 | -8.70 (5.638) | -6.67 (2.517)
  Week 4: number analyzed (Participants) | 9 | 21 | 1 | 5 | 3 | 2 | 1 | 10 | 3
  Week 4 | -2.44 (8.126) | -12.00 (10.277) | 3.00 | -11.20 (10.986) | -15.00 (7.550) | -3.00 (7.071) | -1.00 | -14.40 (7.648) | -14.00 (2.000)
  Week 8: number analyzed (Participants) | 9 | 21 | 1 | 5 | 3 | 2 | 1 | 10 | 3
  Week 8 | -4.22 (6.942) | -17.19 (9.595) | 4.00 | -14.20 (5.020) | -18.67 (10.066) | -2.50 (7.778) | -2.00 | -17.80 (7.540) | -14.00 (4.000)

15. Secondary Outcome: Change From Baseline in CDASI Activity Score at All Scheduled Timepoints Through Week 12 (Stage 3)
Description: The treatment effect was defined as the difference (mean change from baseline at Weeks 1, 4, 8,12 in the active treatment group minus the mean change from baseline at Weeks 1, 4, 8, 12 in the placebo group) in the mean change of CDASI activity score from baseline at scheduled timepoints. The score (range: 0-100) consists of the ES, GHS, PS and AS. ES (range: 0-90) was obtained by summing up scores for the total erythema (ER [0-45], redness of the skin or mucous membranes), scaling (SC [0-30], peeling of the skin) and erosion/ulceration (EU [0-15], presence of the deeper wound). Total ER, SC and EU scores were calculated as a sum of the contributions from 15 individual areas of the body. GHS characterizes papules (swellings) on hand and is a sum of the papule's characterization score (0-6) and ulceration score (0-1). PS (0-2) characterizes abnormalities around nails. The AS (0-1) characterizes hair loss. Higher scores indicate greater disease severity.
Time Frame: Baseline, Week 1, Week 4, Week 8 and Week 12
Population: The Full Analysis Set in Stage 3 (FAS3) included all participants who received at least 1 dose of randomized treatment in Stage 3.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | (Stage 3) Placebo Then Switched to PF-06823859 600 mg IV at Week 12 | (Stage 3) PF-06823859 600 mg IV Then Switched to Placebo at Week 12
Number analyzed (Participants) | 9 | 9
Units on a scale
  Week 1 | -2.00 (3.808) | -2.11 (2.522)
  Week 4 | -3.78 (5.333) | -5.11 (5.555)
  Week 8 | -5.00 (7.382) | -7.78 (6.667)
  Week 12 | -5.89 (8.177) | -8.56 (7.923)

16. Secondary Outcome: Absolute Values of CDASI Activity Score at All Scheduled Timepoints Through Week 12 (All Stages)
Description: The CDASI activity score (range: 0-100) consists of the ES, GHS, PS and AS. ES (range: 0-90) was obtained by summing up scores for the total erythema (ER [0-45], redness of the skin or mucous membranes), scaling (SC [0-30], peeling of the skin) and erosion/ulceration (EU [0-15], presence of the deeper wound). Total ER, SC and EU scores were calculated as a sum of the contributions from 15 individual areas of the body. GHS characterizes papules (swellings) on hand and is a sum of the papule's characterization score (0-6) and ulceration score (0-1). PS (0-2) characterizes abnormalities around nails. The AS (0-1) characterizes hair loss. Higher scores indicate greater disease severity.
Time Frame: Baseline, Week 1, Week 4, Week 8 and Week 12
Population: The FAS included all participants who received at least 1 dose of randomized treatment in any study stage.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | (Stage 1) Placebo | PF-06823859 600 mg IV (Stage 1) | (Stage 2) Placebo | (Stage 2) PF-06823859 150 mg IV | (Stage 2) PF-06823859 600 mg IV | (Amended Stage 2) Placebo Then Switched to PF-06823859 150 mg IV at Week 12 | (Amended Stage 2) Placebo Then Switched to PF-06823859 600 mg IV at Week 12 | (Amended Stage 2) PF-06823859 150 mg IV Then Switched to Placebo at Week 12 | (Amended Stage 2) PF-06823859 600 mg IV Then Switched to Placebo at Week 12 | (Stage 3) Placebo Then Switched to PF-06823859 600 mg IV at Week 12 | (Stage 3) PF-06823859 600 mg IV Then Switched to Placebo at Week 12
Number analyzed (Participants) | 10 | 22 | 1 | 5 | 3 | 2 | 1 | 10 | 3 | 9 | 9
Units on a scale
  Baseline | 31.50 (11.750) | 33.23 (10.323) | 23.00 | 28.60 (9.017) | 37.00 (9.644) | 26.00 (5.657) | 37.00 | 35.40 (13.226) | 30.00 (7.937) | 17.22 (11.595) | 12.56 (8.095)
  Week 1 | 28.90 (12.982) | 27.68 (8.962) | 24.00 | 18.80 (6.535) | 34.67 (9.713) | 19.50 (0.707) | 37.00 | 26.70 (12.667) | 23.33 (9.018) | 15.22 (9.846) | 10.44 (6.894)
  Week 4: number analyzed (Participants) | 9 | 22 | 1 | 5 | 3 | 2 | 1 | 10 | 3 | 9 | 9
  Week 4 | 28.11 (16.136) | 21.23 (11.182) | 26.00 | 17.40 (2.408) | 22.00 (12.490) | 23.00 (1.414) | 36.00 | 21.00 (10.677) | 16.00 (9.539) | 13.44 (8.819) | 7.44 (5.503)
  Week 8: number analyzed (Participants) | 9 | 22 | 1 | 5 | 3 | 2 | 1 | 10 | 3 | 9 | 9
  Week 8 | 26.33 (13.892) | 15.29 (6.157) | 27.00 | 14.40 (5.857) | 18.33 (5.508) | 23.50 (2.121) | 35.00 | 17.60 (10.895) | 16.00 (11.269) | 12.22 (10.883) | 4.78 (4.116)
  Week 12 | 27.11 (14.903) | 12.86 (5.876) | 28.00 | 11.20 (4.817) | 11.00 (3.464) | 23.00 (2.828) | 40.00 | 19.00 (14.087) | 14.67 (9.504) | 11.33 (9.206) | 4.00 (3.464)

17. Secondary Outcome: Absolute Values of CDASI Damage Score at All Scheduled Timepoints Through Week 12 (All Stages)
Description: The Damage Score (DS) was calculated as a sum of the total poilkiloderma score (POLS), total calcinosis score (CALS) and Gotorn's hands damage score (GHDS). The POLS characterizes specific dispigmentation in the particulal area and calcinosis score characterizes calcification of the skin in the particular area. The POLS and the CALS are summed up over 15 individual areas in the body and each of them has range 0-15. The GHDS has the range 0-2 so that the DS has the range 0-32. Higher scores indicate greater disease severity.
Time Frame: Baseline, Week 1, Week 4, Week 8 and Week 12
Population: The FAS included all participants who received at least 1 dose of randomized treatment in any study stage.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | (Stage 1) Placebo | PF-06823859 600 mg IV (Stage 1) | (Stage 2) Placebo | (Stage 2) PF-06823859 150 mg IV | (Stage 2) PF-06823859 600 mg IV | (Amended Stage 2) Placebo Then Switched to PF-06823859 150 mg IV at Week 12 | (Amended Stage 2) Placebo Then Switched to PF-06823859 600 mg IV at Week 12 | (Amended Stage 2) PF-06823859 150 mg IV Then Switched to Placebo at Week 12 | (Amended Stage 2) PF-06823859 600 mg IV Then Switched to Placebo at Week 12 | (Stage 3) Placebo Then Switched to PF-06823859 600 mg IV at Week 12 | (Stage 3) PF-06823859 600 mg IV Then Switched to Placebo at Week 12
Number analyzed (Participants) | 10 | 22 | 1 | 5 | 3 | 2 | 1 | 10 | 3 | 9 | 9
Units on a scale
  Baseline | 4.30 (5.397) | 5.50 (3.901) | 3.00 | 4.20 (3.701) | 7.00 (1.732) | 7.50 (4.950) | 7.00 | 4.70 (4.373) | 7.00 (3.000) | 5.56 (6.044) | 2.00 (1.871)
  Week 1 | 4.90 (5.021) | 5.41 (4.159) | 4.00 | 3.80 (3.347) | 6.33 (3.215) | 6.00 (7.071) | 7.00 | 3.90 (3.542) | 4.67 (2.887) | 6.00 (5.809) | 1.89 (1.764)
  Week 4: number analyzed (Participants) | 9 | 22 | 1 | 5 | 3 | 2 | 1 | 10 | 3 | 9 | 9
  Week 4 | 5.11 (5.278) | 5.23 (3.337) | 4.00 | 3.00 (2.449) | 9.00 (1.732) | 7.00 (5.657) | 7.00 | 4.40 (4.248) | 6.33 (1.528) | 5.22 (4.631) | 1.56 (2.297)
  Week 8: number analyzed (Participants) | 9 | 22 | 1 | 5 | 3 | 2 | 1 | 10 | 3 | 9 | 9
  Week 8 | 5.89 (5.231) | 5.00 (4.427) | 5.00 | 4.40 (2.881) | 8.33 (0.577) | 5.50 (3.536) | 7.00 | 3.70 (3.945) | 4.67 (3.215) | 5.11 (4.859) | 1.00 (1.118)
  Week 12 | 6.33 (5.679) | 5.05 (3.905) | 6.00 | 3.60 (3.286) | 6.33 (1.528) | 4.50 (4.950) | 7.00 | 3.10 (4.358) | 5.00 (1.000) | 5.22 (5.019) | 1.33 (1.581)

18. Secondary Outcome: Absolute Values for Total Improvement Score (TIS) at Week 12 and Intermediate Scheduled Time Points (Stage 3)
Description: The TIS was the sum of all 6 improvement scores where higher score indicates worse status (PhGA [from the MDAAT, 0-20 scale], PtGA [0-10 scale], MMT [0-35 scale], HAQ-DI [0-10 scale], muscle enzymes [0-7.5 scale], and extramuscular global assessment [0-20 scale]) associated with the change in each core set measure. A total improvement score between 0 and 100 corresponded to the degree of improvement, with higher scores corresponding to a greater degree of improvement: of ≥20 represented minimal improvement, a score of ≥40 represented moderate improvement, and a score of ≥60 represented major improvement.
Time Frame: Week 4, Week 8 and Week 12
Population: The FAS3 included all participants who received at least 1 dose of randomized treatment in Stage 3.
Measure: Least Squares Mean (90% Confidence Interval); unit: Units on a scale
Groups:
- Placebo (Stage 3): Participants who were randomized to placebo then PF-06823859 600 mg with a treatment switch at Week 12 in Stage 3.
- PF-06823859 600 mg IV (Stage 3): Participants who were randomized to 600 mg PF-06823859 then placebo with a treatment switch at Week 12 in Stage 3.
Arm/Group | Placebo (Stage 3) | PF-06823859 600 mg IV (Stage 3)
Number analyzed (Participants) | 9 | 9
Units on a scale
  Week 4 | 25.83 [13.15 to 38.52] | 36.67 [23.98 to 49.35]
  Week 8 | 36.67 [23.38 to 49.95] | 49.17 [35.88 to 62.45]
  Week 12 | 36.94 [21.93 to 51.96] | 56.39 [41.38 to 71.40]
Statistical Analysis 1: Comparison: Placebo (Stage 3) vs PF-06823859 600 mg IV (Stage 3); Difference of the active treatment from Placebo at Week 4; Test type: Other; p = 0.1537, Mixed Models Analysis; Least Squares Mean Difference = 10.83, 90% CI 2-sided [-7.10 to 28.77], Standard Error of Mean 10.274
Statistical Analysis 2: Comparison: Placebo (Stage 3) vs PF-06823859 600 mg IV (Stage 3); Difference of the active treatment from Placebo at Week 8; Test type: Other; p = 0.1312, Mixed Models Analysis; Least Squares Mean Difference = 12.50, 90% CI 2-sided [-6.29 to 31.29], Standard Error of Mean 10.761
Statistical Analysis 3: Comparison: Placebo (Stage 3) vs PF-06823859 600 mg IV (Stage 3); Difference of the active treatment from Placebo at Week 12; Test type: Other; p = 0.0647, Mixed Models Analysis; Least Squares Mean Difference = 19.44, 90% CI 2-sided [-1.79 to 40.68], Standard Error of Mean 12.161

19. Secondary Outcome: Change From Baseline in the Core Set Measures (CSM) of the TIS (Global Disease Activity [PhGA] and Extramuscular Global Assessment [EmGA]) (Stage 3)
Description: PhGA: assessment of the severity of disease by the physician. The physician used the visual analog scale and put a mark on 0 cm (best) -10 cm (worst) scale where higher score indicated worse status.
  EmGA: overall evaluation of disease activity in all extramuscular systems using visual analog scale 0 cm (best) -10 cm (worst) scale where higher score indicated worse status.
Time Frame: Baseline, Week 4, Week 8 and Week 12
Population: as for outcome 15
Measure: Least Squares Mean (90% Confidence Interval); unit: Centimeter (cm)
Arm/Group | Placebo (Stage 3) | PF-06823859 600 mg IV (Stage 3)
Number analyzed (Participants) | 9 | 9
Centimeter (cm)
  PhGA Week 4 | -1.00 [-1.89 to -0.11] | -1.68 [-2.57 to -0.79]
  PhGA Week 8 | -1.65 [-2.80 to -0.51] | -2.76 [-3.90 to -1.61]
  PhGA Week 12 | -2.05 [-3.56 to -0.55] | -3.40 [-4.90 to -1.90]
  Extramuscular Global Assessment Week 4 | -1.02 [-2.07 to 0.03] | -1.55 [-2.60 to -0.49]
  Extramuscular Global Assessment Week 8 | -1.91 [-2.80 to -1.01] | -2.48 [-3.38 to -1.58]
  Extramuscular Global Assessment Week 12 | -1.59 [-2.64 to -0.53] | -2.81 [-3.87 to -1.76]

20. Secondary Outcome: Change From Baseline in the CSM of the TIS (PtGA) (Stage 3)
Description: PtGA: assessment of the severity of disease by the participant/participant's guardian, using a visual analog scale from 0 mm (no evidence of disease activity) to 100 mm (extremely active or severe disease activity). Higher score indicated worse status.
Time Frame: Baseline, Week 4, Week 8 and Week 12
Population: The FAS3 included all participants who received at least 1 dose of randomized treatment in Stage 3.
Measure: Least Squares Mean (90% Confidence Interval); unit: Millimeter (mm)
Arm/Group | Placebo (Stage 3) | PF-06823859 600 mg IV (Stage 3)
Number analyzed (Participants) | 9 | 9
Millimeter (mm)
  PtGA Week 4: number analyzed (Participants) | 8 | 9
  PtGA Week 4 | -18.29 [-31.78 to -4.79] | -17.88 [-30.75 to -5.00]
  PtGA Week 8: number analyzed (Participants) | 9 | 8
  PtGA Week 8 | -16.81 [-29.88 to -3.73] | -32.60 [-45.85 to -19.35]
  PtGA Week 12 | -14.04 [-25.91 to -2.17] | -43.81 [-55.68 to -31.95]

21. Secondary Outcome: Change From Baseline in the CSM of the TIS (MMT8 and HAQ01-HAQ-DI) (Stage 3)
Description: Manual Muscle Testing-8 designated muscle groups (MMT-8): was a set of 8 designated muscles tested unilaterally generally on right side (left side used unless right side cannot be used). Potential score range was from 0 to 80, where higher scores denoted better health status.
  HAQ-DI: contained eight sections (including dressing & grooming, arising, eating, walking, hygiene, grip, reach, and activities). Each section had multiple questions that the participant used to rank their functionality and ranged from 0 to 3 where 0 = without any difficulty and 3 = unable to do. For each participant, the average ranking was calculated for each of the eight sections. HAQ-DI had a score range of 0 to 3, where higher score reflected worse status.
Time Frame: Week 4, Week 8 and Week 12
Population: The FAS3 included all participants who received at least 1 dose of randomized treatment in Stage 3.
Measure: Least Squares Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | Placebo (Stage 3) | PF-06823859 600 mg IV (Stage 3)
Number analyzed (Participants) | 9 | 9
Units on a scale
  MMT8 - Derived Week 4 | 7.76 [1.37 to 14.16] | 8.24 [1.84 to 14.63]
  MMT8 - Derived Week 8 | 12.14 [4.60 to 19.68] | 15.24 [7.70 to 22.78]
  MMT8 - Derived Week 12 | 11.65 [2.29 to 21.01] | 21.24 [11.87 to 30.60]
  HAQ01-HAQ-DI Week 4: number analyzed (Participants) | 8 | 9
  HAQ01-HAQ-DI Week 4 | -0.03 [-0.24 to 0.18] | -0.20 [-0.39 to 0.00]
  HAQ01-HAQ-DI Week 8: number analyzed (Participants) | 8 | 9
  HAQ01-HAQ-DI Week 8 | 0.00 [-0.28 to 0.28] | -0.38 [-0.64 to -0.11]
  HAQ01-HAQ-DI Week 12: number analyzed (Participants) | 8 | 9
  HAQ01-HAQ-DI Week 12 | -0.06 [-0.40 to 0.28] | -0.52 [-0.84 to -0.19]

22. Secondary Outcome: Change From Baseline in the CSM of the TIS (Aldolase and Creatine Kinase) (Stage 3)
Description: The LS mean (with 90% CI) of CSM of the TIS (aldolase and creatine kinase) at weeks 4, 8, 12 were presented.
Time Frame: Baseline, Week 4, Week 8 and Week 12
Population: The FAS3 included all participants who received at least 1 dose of randomized treatment in Stage 3.
Measure: Least Squares Mean (90% Confidence Interval); unit: Units per litre (U/L)
Arm/Group | Placebo (Stage 3) | PF-06823859 600 mg IV (Stage 3)
Number analyzed (Participants) | 9 | 9
Units per litre (U/L)
  Aldolase Week 4: number analyzed (Participants) | 9 | 8
  Aldolase Week 4 | -0.19 [-1.34 to 0.96] | -3.09 [-4.25 to -1.92]
  Aldolase Week 8: number analyzed (Participants) | 9 | 7
  Aldolase Week 8 | -1.31 [-2.45 to -0.16] | -3.57 [-4.74 to -2.40]
  Aldolase Week 12: number analyzed (Participants) | 8 | 7
  Aldolase Week 12 | -0.66 [-2.18 to 0.86] | -3.20 [-4.76 to -1.64]
  Creatine Kinase Week 4 | -37.96 [-119.16 to 43.24] | -157.48 [-238.68 to -76.28]
  Creatine Kinase Week 8 | -70.96 [-137.03 to -4.90] | -175.93 [-241.99 to -109.86]
  Creatine Kinase ) Week 12: number analyzed (Participants) | 9 | 8
  Creatine Kinase ) Week 12 | -39.85 [-125.71 to 46.01] | -185.77 [-273.92 to -97.62]

ADVERSE EVENTS:
Time Frame: Up to Week 40
Description: The safety analysis set includes all participants who received at least one dose of randomized treatment in any stage. The AEs reported were treatment emergent.
Groups:
- Placebo: Participants who received placebo in any stage.
- PF-06823859 150 mg IV: Participants who received PF-06823859 150 mg IV in any stage.
- PF-06823859 600 mg IV: Participants who received PF-06823859 600 mg IV in any stage.
- Total: This arm included all participants (32, 9, 16 and 18 participants who were randomized and treated in Stage 1, Stage 2, Amended Stage 2, and Stage 3, respectively) in the safety analysis set
Arm/Group | Placebo | PF-06823859 150 mg IV | PF-06823859 600 mg IV | Total
All-Cause Mortality (participants affected / at risk) | 1/45 | 0/17 | 1/47 | 1/75
Serious Adverse Events (participants affected / at risk) | 3/45 | 0/17 | 4/47 | 5/75
Other Adverse Events (participants affected / at risk) | 22/45 | 13/17 | 18/47 | 45/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=45) | PF-06823859 150 mg IV (N=17) | PF-06823859 600 mg IV (N=47) | Total (N=75)
Cytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1
Colitis microscopic (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Ocular icterus (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Central nervous system lesion (Nervous system disorders) | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=45) | PF-06823859 150 mg IV (N=17) | PF-06823859 600 mg IV (N=47) | Total (N=75)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 3 | 4
Nausea (Gastrointestinal disorders) | 2 | 0 | 3 | 5
Fatigue (General disorders) | 4 | 1 | 1 | 6
Sinusitis (Infections and infestations) | 3 | 1 | 0 | 4
Tooth abscess (Infections and infestations) | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 4 | 5
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 2
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Blood potassium decreased (Investigations) | 0 | 1 | 1 | 2
SARS-CoV-2 test positive (Investigations) | 4 | 0 | 1 | 4
Weight increased (Investigations) | 1 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 7 | 3 | 6 | 15
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 1
Mental impairment (Nervous system disorders) | 0 | 1 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 1 | 1 | 6
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-09-20): https://cdn.clinicaltrials.gov/large-docs/93/NCT03181893/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-09): https://cdn.clinicaltrials.gov/large-docs/93/NCT03181893/SAP_001.pdf